CLINICAL TRIAL: NCT00532714
Title: Phase II Study of Irinotecan Plus Capecitabine in Patients With Antracycline and Taxane Pretreated Metastatic Breast Cancer
Brief Title: Phase II Study of Irinotecan/Capecitabine in Patients With Antracycline/Taxane Pretreated MBC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Center, Korea (Other Government)
Responsible Party: Principal Investigator, Jungsil Ro, Chief, Center for Clinical Trials, National Cancer Center, Korea, National Cancer Center, Korea
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCCCTS-06-201
Record Dates: First submitted 2007-09-19; First posted 2007-09-20 (Estimated); Last update posted 2011-12-30 (Estimated); Status verified 2011-12

CONDITIONS: Breast Cancer Metastatic
MeSH Terms: interventions — Irinotecan; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Irinotecan plus capecitabine (No Intervention): Irinotecan 80 mg/m2 (intravenously once a week for 2 weeks (Days 1 and 8) followed by 1-week rest period) Capecitabine (orally at a dose of 1,000 mg/m2 twice daily 3-week cycles (2 weeks of treatment followed by a 1-week rest period))
  Interventions: Drug: Irinotecan plus capecitabine

INTERVENTIONS:
Drug: Irinotecan plus capecitabine — Irinotecan 80 mg/m2 intravenously for 90 minutes once a week for 2 weeks (Days 1 and 8) followed by 1-week rest period.
  Capecitabine is administered orally at a dose of 1,000 mg/m2 twice daily (total daily dose 2,000 mg/m2) as an intermittent regimen in 3-week cycles (2 weeks of treatment followed by a 1-week rest period).
  Other Names: Crabcan; Xeloda

SUMMARY:
To evaluate the response rate of capecitabine and irinotecan combination therapy in patients with metastatic breast cancer

DETAILED DESCRIPTION:
This is a nonrandomized, open-label, phase II study of irinotecan plus capecitabine in patients with metastatic breast cancer previously treated with anthracyclines and taxanes. Up to 44 qualified patients will be enrolled according to the exact single stage design.

Irinotecan 90 mg/m2 intravenously for 90 minutes once a week for 2 weeks (Days 1 and 8) followed by 1-week rest period. Capecitabine is administered orally at a dose of 1,000 mg/m2 twice daily (total daily dose 2,000 mg/m2) as an intermittent regimen in 3-week cycles (2 weeks of treatment followed by a 1-week rest period). For practical reasons, capecitabine doses are rounded to the nearest dose that could be administered with a combination of 500-mg and 150-mg tablets of drug. Capecitabine is given approximately 12 hours apart and taken orally with water within 30 minutes after ingestion of food (breakfast or dinner).

ELIGIBILITY:
Inclusion Criteria:

* Histologic or cytologic diagnosis of breast cancer Stage IV or recurrent.
* Previous chemotherapy with anthracyclines and taxane in adjuvant setting
* Previous hormonal therapy in adjuvant and metastatic setting is allowed
* Prior radiation therapy is allowed as long as the irradiated area is not the only source of measurable disease.
* No other forms of cancer therapy, such as radiation, immunotherapy for at least 3 weeks before the enrollment in study.
* Performance status of 0, 1, 2 on the ECOG criteria.
* Clinically measurable disease, defined as uni-dimensionally measurable lesions with clearly defined margins on x-ray, CT scan, MRI or physical examination. Lesions serving as measurable disease must be at least 1 cm, as defined by x-ray, CT scan, MRI, or physical examination.
* Estimated life expectancy of at least 12 weeks.
* Patient compliance that allow adequate follow-up.
* Adequate hematologic (WBC count ³ 3,000/mm3, platelet count ³ 100,000/mm3), hepatic (bilirubin level £ 1.5 mg/dL), and renal (creatinine concentration £ 1.5 mg/dL) function.
* Informed consent from patient or patient's relative.
* Males or females at least 18 years of age.
* If female: childbearing women should use non-hormonal contraceptive method

Exclusion Criteria:

* MI within preceding 6 months or symptomatic heart disease, including unstable angina, congestive heart failure or uncontrolled arrhythmia.
* Serious concomitant infection.
* Second primary malignancy (except in situ carcinoma of the cervix or adequately treated basal cell carcinoma of the skin or prior malignancy treated more than 5 years ago without recurrence).

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2006-08; Primary Completion 2008-04 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
To evaluate the response rate of capecitabine and irinotecan combination therapy in patients with metastatic breast cancer | 2009

SECONDARY OUTCOMES:
To investigate the toxicity profiles of capecitabine and irinotecan combination To determine time to progression and overall survival | 2009

CONTACTS AND LOCATIONS:
Overall Officials: Jungsil Ro, M.D., Principal Investigator — National Cancer Center
Locations (1):
- National Cancer Center, 809 Madu1-dong, Ilsandong-gu, Goyang-si, Gyeonggi-do, South Korea